CLINICAL TRIAL: NCT01022645
Title: Postpartum Glucose Tolerance in Women With Recent Gestational Diabetes Using the Levonorgestrel IUD and Non-Hormonal Contraception: A Prospective Cohort Study
Brief Title: Postpartum Glucose Tolerance With Levonorgesterel IUD Use in Women With Recent Gestational Diabetes
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Jessica Kiley, Prinicipal Investigator, Northwestern University
Other Study IDs: STU00014472; SFP3-3
Record Dates: First submitted 2009-11-25; First posted 2009-12-01 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Gestational Diabetes; Glucose Intolerance; Type 2 Diabetes; Intrauterine Contraception
Keywords: Intrauterine device; Gestational diabetes; Postpartum contraception; Postpartum birth control
MeSH Terms: conditions — Diabetes, Gestational; Glucose Intolerance; Diabetes Mellitus, Type 2 | interventions — Sterilization, Tubal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Levonorgestrel IUD
  Interventions: Device: Mirena (Levonorgestrel IUD)
- Copper IUD or Tubal Ligation
  Interventions: Device: Paragard (Copper IUD ) or Tubal Ligation

INTERVENTIONS:
Device: Mirena (Levonorgestrel IUD) — Release of intrauterine levonorgestrel for contraception, approved for up to 5 years' use
  Other Names: Mirena IUD
  Groups: Levonorgestrel IUD
Device: Paragard (Copper IUD ) or Tubal Ligation — Copper IUD placed to provide contraception for up to 10 years
  Other Names: Paragard IUD
  Groups: Copper IUD or Tubal Ligation

SUMMARY:
The study is being done in order to gain information on the most suitable types of birth control in women who recently had gestational diabetes, or diabetes diagnosed during pregnancy. The intrauterine device (IUD) is a highly effective form of birth control. It is inserted into the uterus and prevents pregnancy for either 5 or 10 years, depending on the type of IUD (hormone-releasing or copper). The hormone-releasing IUD works for 5 years and releases a hormone called a progestin into the uterus. The copper IUD contains no hormones and works for 10 years. The IUD is an excellent form of birth control postpartum, but it is unknown if the hormone-releasing IUD will affect blood sugars and increase a woman's risk of becoming diabetic when she's not pregnant. The hypothesis is that the hormone-containing IUD will NOT increase blood sugars, so women who use the hormone-containing IUD will have similar blood sugars to those who use the copper IUD or have had their tubes tied (no hormones).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years at the time of enrollment
2. Single gestation in the current pregnancy
3. GDM in the current pregnancy, diagnosed by 2- or 3-hour oral glucose tolerance test (OGTT) performed at 24-32 weeks gestation
4. Desires intrauterine contraception or tubal ligation postpartum
5. Willing and able to read and sign an informed consent form in English
6. Willing to comply with the study protocol

Exclusion Criteria:

1. History of pre-gestational DM, type 1 or 2
2. Pregnancy conceived with assisted reproductive technologies
3. Positive for human immunodeficiency virus (HIV) infection
4. Desires repeat pregnancy within the first 12 months following delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Postpartum women with gestational diabetes in the last pregnancy
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2009-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance at 12 months postpartum. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jessica W Kiley, MD, MPH, Principal Investigator — Northwestern Universeity
Locations (1):
- Northwestern Medical Faculty Foundation; Northwestern Memorial Hospital, Chicago, Illinois, United States